CLINICAL TRIAL: NCT07071025
Title: Preventing Perinatal Anxiety: Testing an Internet-delivered Intervention
Acronym: P-POD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: University of Vermont (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle Roley-Roberts, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2210663965; R15HD109689 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Disorder
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventing Postpartum Onset Distress (P-POD) (Experimental): P-POD is an online self-guided program designed to reduce and prevent perinatal anxiety in at-risk women in West Virginia.
  Interventions: Behavioral: Preventing Postpartum Onset Distress (P-POD)
- Anxiety Education (ANX-ED) (Placebo Comparator): ANX-ED will be adapted from an already-established in-person anxiety education control condition and will be modified to an Internet-based, self-guided program that serves as an attention control to P-POD.
  Interventions: Behavioral: Anxiety Education (ANX-ED)

INTERVENTIONS:
Behavioral: Preventing Postpartum Onset Distress (P-POD) — P-POD contains ten interactive and didactic modules lasting approximately 30 minutes each. Seven mother-directed modules are designed to educate pregnant women about perinatal anxiety (psychoeducation), teach women to change their thinking patterns (cognitive restructuring), and guide women through testing their dysfunctional beliefs and fears (behavioral experiments). Each of these modules engage the pregnant woman in various self-guided exercises to consolidate the lessons learned. In addition, three partner-directed modules are designed to educate partners about perinatal anxiety, coach partners on providing emotional and social supports to pregnant women at risk for perinatal anxiety, and prepare partners for developmentally normative changes in their relationships following birth. Modules are designed to be completed weekly during the second trimester.
  Arms: Preventing Postpartum Onset Distress (P-POD)
Behavioral: Anxiety Education (ANX-ED) — ANX-ED educates women and their partners about seven anxiety and related disorders. ANX-ED contains ten interactive and didactic modules lasting approximately 30 minutes each. Seven mother-directed modules and three partner-directed modules will educate participants about generalized anxiety disorder, social anxiety disorder, panic disorder, specific phobia, obsessive-compulsive disorder, and posttraumatic stress disorder. Specifically, modules will include the diagnostic criteria, prevalence, and etiology of the disorders. They will also include animated examples of mothers experiencing the disorders described in each module. Each module engages the pregnant woman (or partner) in various self-guided exercises to consolidate the material learned.
  Arms: Anxiety Education (ANX-ED)

SUMMARY:
Postpartum anxiety disorders are the most prevalent postpartum psychiatric conditions. The purpose of this study is to evaluate the Internet-delivered postpartum anxiety and obsessive-compulsive disorder (OCD) prevention program, called "Preventing Postpartum Onset Distress", or P-POD. The overarching goal of this study is to conduct a randomized control trial of P-POD, an online program designed to reduce and prevent perinatal anxiety in at-risk women in West Virginia. Investigators will test the effects of P-POD compared to an anxiety education control intervention on risk factors for perinatal anxiety and assess mothers' anxiety symptoms, relationships with their partners, and relationships with their infants at 8-weeks postpartum. Eligible women and their partners will be consented at the start of the second trimester of pregnancy. Couples will be randomized into either the P-POD (active) or ANX-ED (control) intervention. Couples will then begin to work through the ten intervention modules: seven modules for women, at a recommended rate of one per week, and three modules for partners, at a recommended rate of no more than one per week. Women will complete brief weekly phone "coaching calls" to encourage module completion, ensure understanding of material, and answer any content-related or technical questions. Ten weeks after the pre-intervention assessment, women will complete the post-intervention assessment (same measures as pre-assessment).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and entering second trimester
* In a romantic relationship
* Partner must be agreeable to participate
* State Trait Anxiety Inventory-Trait Total ≥ 44 and/or Obsessive Beliefs Questionnaire-44 Total ≥ 139

Exclusion Criteria:

-Must speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant individuals
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory-Trait (STAI-Trait) | Change from Baseline to Week 10
  Change in STAI-Trait score. This is a 20-item self-report used to assess dispositional levels of anxiety. It is widely used, sensitive to treatment, has strong psychometric properties, and includes items that would be relevant to pregnant women. The STAI-Trait Total Score will be used before and after P-POD to assess change in prenatal trait anxiety. The STAI-Trait total score ranges from 20 to 80. Higher numbers represent more anxiety (worse outcome).
Change in Obsessive Beliefs Questionnaire (OBQ) | Change from Baseline to Week 10
  Change in Obsessive Beliefs Questionnaire (OBQ) score. This measure assesses dysfunctional beliefs related to OCD in 44 items on a 7-point Likert-type scale, with items summed; higher scores indicate more dysfunctional beliefs. The OBQ has strong psychometric properties and has demonstrated sensitivity to treatment with pregnant women.

SECONDARY OUTCOMES:
Change in Perinatal Interpretations Questionnaire (PIQ) | Change from Baseline to Week 10
  The PIQ will be administered to assess change in negative interpretations. This measure asks participants to read and imagine themselves in two scenarios (e.g., not checking on baby while he/she sleeps) and then rate the likelihood of eight interpretations related to each scenario (e.g., "your baby is not safe") on a 5-point Likert-type response scale. The 16 items are summed, higher scores indicate more negative perinatal interpretations.
Change in Social Provisions Checklist (SPC) | Change from Baseline to 8-weeks postpartum
  The SPC will be administered to assess change in partner support. This measure asks participants to rate the extent to which they receive different benefits (e.g., emotional closeness) from their romantic partner. It consists of 30 items on a 5-point Likert-type scale; items are summed and higher scores indicate more perceived support. The SPC has strong internal reliability and construct validity.
Overall Anxiety Severity and Impairment Scale (OASIS) | 8-weeks postpartum
  The OASIS will be administered to assess severity of postpartum anxiety. This 5-item self-report of anxiety symptom severity and impairment has strong reliability, convergent validity, and discriminant validity in both nonclinical and clinical samples, is sensitive to treatment and has been used with perinatal women. Items are scored on a 5-point scale and summed; higher scores are indicative of higher symptom severity and impairment.
Dimensional Obsessive-Compulsive Scale (DOCS) | 8-weeks postpartum
  The DOCS will be administered to assess severity of postpartum OCD symptoms. This 20-item self-report of OCD symptom severity has good internal consistency, construct validity, discriminant validity, and sensitivity to treatment, and has been recommended for use in pregnant women. Items are rated on a 5-point Likert-type scale and are summed; higher numbers are indicative of higher symptom severity.
Edinburgh Postpartum Depression Scale (EPDS) | 8-weeks postpartum
  The EPDS will be administered to assess severity of postpartum depression. This 10-item screening tool assesses postpartum depression symptoms in perinatal women and has shown strong evidence for validity and reliability. Items are scored on a 4-point scale and summed; higher scores indicate higher severity of depression symptoms.
Couple Satisfaction Index-4 (CSI-4) | 8-weeks postpartum
  The CSI-4 will be administered to assess relationship satisfaction of both the woman and partner. This index assesses satisfaction in relationships through one item with a 6-point Likert scale and three items with a 5-point Likert scale. Strong reliability, construct validity, and convergent validity has been demonstrated. The CSI-4 items are summed, with higher numbers suggesting more relationship satisfaction.
Postpartum Bonding Questionnaire (PBQ) | 8-weeks postpartum
  The PBQ will be administered to assess mother-infant bonding. This measure contains 25 items assessing maternal perceptions of bonding with their infant on a 6-point Likert-type scale. It includes the following subscales: impaired bonding, rejection and pathological anger, infant-focused anxiety, incipient abuse. The PBQ has strong reliability and has good concurrent validity with maternal mental health indicators.
Five Minute Speech Sample (FMSS) | 8-weeks postpartum
  Participants are recorded (via Zoom). The participant is given the following instructions: "I'd like to hear your thoughts about [baby's name] in your own words and without my interrupting you with any questions or comments. When I ask you to begin, I'd like you to speak for 5 minutes, telling me what kind of a baby [baby's name] is and how the two of you get along together. After you have begun to speak, I prefer not to answer any questions. Are there any questions you would like to ask me before we begin?". The recording is coded by 2 independent research assistants. Researchers code for the following categories of statements: quality of initial statement, quality of relationship with baby, emotional over-involvement, and criticism. A randomly selected 20% of recordings will be double coded to assess interrater reliability.
Qualitative Interview | 8-weeks postpartum
  We will use a Qualitative Description approach, which results in a rich description of experiences or perceptions of participants, using language from the collected data through low-inference (or data-near) interpretations during data analysis. We plan to interview approximately 50 women (25 per condition), though we will code interviews in batches and stop recruitment following thematic saturation. Content analysis (inductive approach) will be used to systematically reduce data into coded units that are clustered into categories according to shared characteristics. Qualitative data analysis software (NVivo 12) will be used for data management and coding purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Roley Roberts, PhD, Principal Investigator — West Virginia University
Locations (1):
- Life Sciences Building, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No